CLINICAL TRIAL: NCT05112250
Title: Intravascular Lithotripsy for the Treatment of Stent Underexpansion: the Multicenter IVL-DRAGON Registry
Brief Title: IVL for Stent Underexpantsion
Acronym: IVL-DRAGON
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Collaborators: Wojciech Wojakowski (Unknown)
Responsible Party: Principal Investigator, Wojciech Wańha, Associate professor, Medical University of Silesia
Other Study IDs: 06
Record Dates: First submitted 2021-10-19; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: In Stent Restenosis; Coronary Artery Calcification; Intravascular Lithotripsy
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Percutaneous Coronary Intervention — Intravascular lithotripsy (IVL)

SUMMARY:
The IVL-Dragon Registry was a multicenter study that enrolled consecutive patients with stent underexpansion treated with IVL in high-volume PCI centers. The primary efficacy endpoint was clinical success, defined as a reduction of stent underexpansion to <30% with no evidence of in-hospital device-oriented composite end point (DOCE) (defined as a composite of cardiac death, target lesion revascularization, and target vessel myocardial infarction).

ELIGIBILITY:
Inclusion Criteria:

* stent underexpansion treated with intravascular lithotripsy (IVL)

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients with stent underexpansion treated with intravascular lithotripsy (IVL)
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 30 days
  Reduction of stent underexpansion to the value of <30% with no evidence of in-hospital device-oriented composite end point (DOCE)

SECONDARY OUTCOMES:
DOCE | 30 days
  composite of cardiac death, target lesion revascularization (TLR), target lesion revascularization, (TLR), and target vessel myocardial infarction (MI)

CONTACTS AND LOCATIONS:
Locations (16):
- Poland (16):
  - Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok
  - First Department of Cardiology, Medical University of Gdansk, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow
  - Miedziowe Centrum Zdrowia S.A., Lubin
  - Department of Cardiology, University Hospital, Institute of Medical Sciences, Opole
  - Department of Cardiology, Poznan University of Medical Sciences, Poznan
  - Department of Cardiology, Poznan
  - Department of Cardiology, The Ministry of Internal Affairs and Administration Hospital, Rzeszow, Rzeszów
  - 1st Department of Cardiology, Medical University of Warsaw, Warsaw
  - Department of Cardiology and Internal Diseases, Military Institute of Medicine, Warsaw
  - Department of Interventional Cardiology and Angiology, National Institute of Cardiology, Warsaw, Poland, Warsaw
  - Department of Invasive Cardiology, Centre of Postgraduate Medical Education, Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Department of Invasive Cardiology, Wejherowo, Wejherowo
  - Centre for Heart Disease, University Hospital Wroclaw Department of Heart Disease, Wroclaw Medical University, Wroclaw
  - Third Department of Cardiology, Medical University of Katowice, Zabrze

IPD SHARING:
Plan to Share IPD: Undecided